CLINICAL TRIAL: NCT04748094
Title: Quantification of Abdominal Organ Motion Using Magnetic Resonance Imaging (MRI)
Brief Title: Quantification of Abdominal Organ Motion Using MRI
Acronym: QUANTUM
Status: Completed | Type: Observational
Sponsor: The Christie NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: CFTSp166
Record Dates: First submitted 2021-01-27; First posted 2021-02-10 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2025-08

CONDITIONS: Cancer
Keywords: MRI
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Free-breathing versus Compression: This cohort of volunteers and patients will undergo imaging on the MR-Linac investigating free-breathing motion, and comparing it to motion using an abdominal compression device.
  Interventions: Device: Compression belt
- Free-breathing versus Breath-holding: This cohort of volunteers and patients will undergo imaging on the MRSim investigating free-breathing motion and comparing it to visually-guided breath-hold motion (and reproducibility).
  Interventions: Other: Visual Guided Breath-hold

INTERVENTIONS:
Device: Compression belt — The abdominal belt is fastened around the lower abdomen and inflated (like an inner tube) to apply pressure to the belly and reduce the motion associated with respiration (breathing)
  Groups: Free-breathing versus Compression
Other: Visual Guided Breath-hold — A small tracer will be place on the lower abdomen that will feedback to a computer screen that will have graphics to show you if the participant is in breath-hold or not.
  Groups: Free-breathing versus Breath-holding

SUMMARY:
The primary aim of the study is to quantify abdominal motion in order to optimise MR imaging. The study will compare three-motion management strategies a) free-breathing, b) using an abdominal compression belt and c) using MRI-compatible visually guided breath-holds.

ELIGIBILITY:
Inclusion Criteria:

Healthy volunteers

* 18 years or older,
* no MRI contra-indications
* must agree to registration as a non-patient in CWP (the local electronic healthcare records system) and have their MRIs read and reviewed for incidental findings by a clinical radiologist

Patient Volunteers

* undergoing radiotherapy to the abdominal region at the Christie NHS Foundation Trust
* Over 18 years of age

Exclusion Criteria:

* Any contraindications to MRI identified after MRI safety screening including completion of an MRI Safety Screening Form
* Unable to tolerate MRI scan
* Pregnancy
* Colostomy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients or staff at The Christie NHS Foundation Trust
Sampling Method: Non-Probability Sample
Enrollment: 23 (Actual)
Dates: Start 2021-05-21 (Actual); Primary Completion 2023-03-15 (Actual); Study Completion 2023-03-15 (Actual)

PRIMARY OUTCOMES:
MRI Motion Management SOP | through study completion, approximately 6 months
  Development and implementation of an MRI protocol suitable for organ motion characterisation for the abdomen. Determination of the benefit of motion management strategies for abdominal radiotherapy.

SECONDARY OUTCOMES:
Quantification of motion | through study completion, approximately 6 months
  Quantification of intra-abdominal inter and intra-fraction motion with and without abdominal compression and visually guided breath holds using MR imaging. Comparative analysis of comparable treatment plans with and without abdominal compression and visually guided breath holds on relevant treatment planning software for PBT and MRL. Development of process to evaluate patient compliance when using a commercial available abdominal compression belt and visually guided breath-hold.

CONTACTS AND LOCATIONS:
Locations (1):
- The Christie NHS Foundation Trust, Manchester, Greater Manchester, United Kingdom